CLINICAL TRIAL: NCT03619460
Title: Clinical Efficacy of a New Piezoelectric Technique for Wisdom Teeth Extraction Without Using Manual Tools: a Clinical Randomized Controlled Study.
Brief Title: Clinical Efficacy of a New Piezoelectric Technique for Wisdom Teeth Extraction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Azienda Ospedaliera di Bolzano (Other)
Responsible Party: Principal Investigator, Grusovin Maria Gabriella, Principal investigator, Azienda Ospedaliera di Bolzano
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0060125-BZ
Record Dates: First submitted 2018-07-20; First posted 2018-08-08 (Actual); Last update posted 2019-01-11 (Actual); Status verified 2019-01

CONDITIONS: Impacted Third Molar Tooth
Keywords: wisdom teeth; extraction; piezoelectric technique

STUDY DESIGN:
Intervention Model Description: All patients will take amoxicillin + clavulanic acid and Ibuprofen 600mg . Mepivacain with 1:100.000 adrenalin will be used for anesthesia. Local infiltration of Desamethasone 4mg and intraoral disinfection of the surgical area with povidone iodine will be done.
  A full thickness flap will be raised after a sulcular incision from the mesial buccal aspect of the second molar to the distal aspect of the third one where a releasing incision begins describing an open V shape.
  In the Piezoelectric group Piezoelectric tools will be used. In the conventional group manual tools and burs with a straight handpiece will be used. The flap will be sutured using a 3/0 suture. Levobupivacaine hydrochloride 5mg will be injected at the end of the procedure in the site of the operation
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Sequentially sealed opaque envelopes will be opened by a nurse not involved in the treatment of the patient and a number will be assigned to the patients included in the study. The randomization code will be disclosed at the end of the statistical analysis. The doctor who will evaluate the complications, the duration of the procedure and the healing will be not aware of the type of treatment provided to the patients, nor will be the patients.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- piezoelectric extraction (Experimental): The flap will be raised using a Piezoelectric elevator, the eventual bone around the third molar crown will be removed with the same piezoelectric lever used for luxation and root extraction. The eventual rizectomy will be performed using a piezoelectric saw.
  Interventions: Procedure: piezoelectric extraction
- conventional extraction (Active Comparator): The flap will be raised using a manual elevator and the eventual bone around the third molar crown will be removed with a bone bur with a straight handpiece while the eventual rizectomy will be performed using a bone bur. Manual levers will be used for luxation and tooth extraction
  Interventions: Procedure: conventional extraction

INTERVENTIONS:
Procedure: piezoelectric extraction — Only Piezoelectric device will be used for surgical wisdom teeth extraction
  Arms: piezoelectric extraction
Procedure: conventional extraction — Only manual instruments and burs on straight handpick will be used for wisdom teeth extraction
  Arms: conventional extraction

SUMMARY:
the aim of this randomized controlled clinical study is to evaluate the efficacy of a new piezoelectric technique for wisdom teeth extraction without using manual tools versus the conventional one.Patients referred to the hospital of Bolzano for wisdom tooth extraction will be randomly divided in two groups. In the test group all the procedure will be performed using piezoelectric instruments, while in the control one conventional manual instruments will be used. Main outcome measures are patient pain and complications, secondary outcome measures are duration of the surgical treatment and soft tissue healing

DETAILED DESCRIPTION:
Wisdom teeth extraction can be difficult and patient can suffer post operative swelling and pain. A new piezoelectric technique for wisdom teeth extraction was developed and it showed promising results in terms of surgical effectiveness and patients post operative complications. The aim of the study is to compare the new technique with special designed piezoelectric tools with the traditional one in a randomized controlled way. The same procedures are to be followed for teeth extraction except for the use of a piezoelectric lever in one group and a manual lever in the other one. The study is a mono-center, pragmatic, randomised clinical trial (RCT) of parallel group design. The trial would have one week follow up. All patients referred to the Dental Department of S.Maurizio Hospital (Bolzano, Italy) for the extraction of wisdom teeth are considered eligible for the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients referred for wisdom tooth extraction
* Patients older than 18 years old and able to sign the informed consent

Exclusion Criteria:

* General contraindications to surgery.
* Patients irradiated in the head and neck area.
* Immunosuppressed or immunocompromised patients.
* Patients who took or are taking bisphosphonates intravenously.
* Uncontrolled diabetes
* Presence of oral pathologies that seriously involved oral mucosa
* Patients with poor oral hygiene and motivation.
* Patients with oral pathologies with serious mucosal involvement
* Pregnancy or lactation.
* Addiction to alcohol or drugs.
* Psychiatric problems.
* Patients with an acute infection inflammation around the tooth to be extracted.
* Wisdom teeth with roots attached or positioned around the nerve
* Patients unable to come to the required follow up visits

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-03-01 (Estimated); Study Completion 2019-03-01 (Estimated)

PRIMARY OUTCOMES:
Subjective Patient's perception of pain | 7 days
  - a visual analogue scale with categorical value from 0 to 10 will be filled by the patient at 6 hours after surgical treatment and every morning in the following 7 days.

SECONDARY OUTCOMES:
Patient's perception of pain | 7 days
  the number of analgesics taken by the patients will be recorded: the patient will register the number of tablets taken after the surgery up to the 7th day
Duration of the surgical treatment | 1 day
  measured from opening of the flap to end of the extraction, suturing excluded
Complication | 7 days
  Any intrasurgical complication will be registered. Besides swelling and trismus will be evaluated at half an hour, 3 and 7 days after the surgery. Bleeding will be evaluated half an hour after the treatment.
Healing of soft tissues | 7 days
  presence of normal healing, inflammation, suppuration will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: FABRIZIO FONTANELLA, MDS, Study Director — BOLZANO HOSPITAL
Locations (1):
- Bolzano Hospital, Bolzano, Italy

IPD SHARING:
Plan to Share IPD: Undecided
CLINICAL STUDY REPORT

REFERENCES:
- [Background] Piersanti L, Dilorenzo M, Monaco G, Marchetti C. Piezosurgery or conventional rotatory instruments for inferior third molar extractions? J Oral Maxillofac Surg. 2014 Sep;72(9):1647-52. doi: 10.1016/j.joms.2014.04.032. Epub 2014 May 6. PMID 25109581
- [Background] Vercellotti T Cap. 4 Tecniche di Estrazione dentale pag 31- 47 Piezosurgery elementi essenziali. Ed Quintessenza 2009
- [Background] Vercellotti T Cap.8 Nuove tecniche estrazioni dentali pag. 185 -255. La chirurgia ossea piezoelettrica: una nuova era. Ed Quintessenza 2016
- [Result] Barone A, Marconcini S, Giacomelli L, Rispoli L, Calvo JL, Covani U. A randomized clinical evaluation of ultrasound bone surgery versus traditional rotary instruments in lower third molar extraction. J Oral Maxillofac Surg. 2010 Feb;68(2):330-6. doi: 10.1016/j.joms.2009.03.053. Epub 2010 Jan 15. PMID 20116704
- [Result] Itro A, Lupo G, Marra A, Carotenuto A, Cocozza E, Filipi M, D'Amato S. The piezoelectric osteotomy technique compared to the one with rotary instruments in the surgery of included third molars. A clinical study. Minerva Stomatol. 2012 Jun;61(6):247-53. English, Spanish. PMID 22669054
- [Result] Goyal M, Marya K, Jhamb A, Chawla S, Sonoo PR, Singh V, Aggarwal A. Comparative evaluation of surgical outcome after removal of impacted mandibular third molars using a Piezotome or a conventional handpiece: a prospective study. Br J Oral Maxillofac Surg. 2012 Sep;50(6):556-61. doi: 10.1016/j.bjoms.2011.10.010. Epub 2011 Nov 15. PMID 22088359
- [Result] Sortino F, Pedulla E, Masoli V. The piezoelectric and rotatory osteotomy technique in impacted third molar surgery: comparison of postoperative recovery. J Oral Maxillofac Surg. 2008 Dec;66(12):2444-8. doi: 10.1016/j.joms.2008.06.004. PMID 19022121
- [Result] Spinato S, Rebaudi A, Bernardello F, Bertoldi C, Zaffe D. Piezosurgical treatment of crestal bone: quantitative comparison of post-extractive socket outcomes with those of traditional treatment. Clin Oral Implants Res. 2016 Mar;27(3):361-6. doi: 10.1111/clr.12555. Epub 2015 Jan 30. PMID 25639687
- [Result] Vercellotti T. Technological characteristics and clinical indications of piezoelectric bone surgery. Minerva Stomatol. 2004 May;53(5):207-14. English, Italian. PMID 15263877